CLINICAL TRIAL: NCT02778672
Title: Thermal Imaging of the Lung on a Smartphone to Differentiate Bacterial From Non Bacterial Causes of Pneumonia
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Patricia Hibberd, Chair School of Public Health, Department of Global Health, Boston University
Other Study IDs: H-35690; OPP1140544 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Pneumonia, Bacterial; Infections, Bacterial
Keywords: bacterial pneumonia; children; diagnosing pneumonia; thermal imaging
MeSH Terms: conditions — Pneumonia, Bacterial; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants with potential pneumonia
  Interventions: Other: Thermal imaging of infant's chest with a mobile phone

INTERVENTIONS:
Other: Thermal imaging of infant's chest with a mobile phone

SUMMARY:
This is a study of up to 275 participants from birth to 12 months who are having a chest x-ray while a patient at the Queen Elizabeth Central Hospital in Blantyre, Malawi. Participants will have thermal pictures of their chest taken by trained study staff using a Smartphone and a FLIR ONE attachment. Thermal images will be read by trained study staff to determine if bacterial pneumonia is present. Results of the thermal images will then be compared to the results of the chest X-ray. If additional images of the chest are available, additional thermal images will be taken of the same location within 24 hours of the other image.

ELIGIBILITY:
Inclusion Criteria:

* patient at Queen Elizabeth Central Hospital in Blantyre, Malawi
* having chest x-ray done to rule out pneumonia
* thermal image can be taken within 24 hours of chest x-ray
* parent/guardian provides written informed consent

Exclusion Criteria:

* none

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 275 Infants at Queen Elizabeth Central Hospital in Blantyre, Malawi having a chest x-ray done to rule out pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Rate of concordance between thermal image and the concurrent chest x-ray regarding the diagnosis of bacterial pneumonia | Within 24 hours of the chest x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Hibberd, MD, PhD, Principal Investigator — Boston University
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No